CLINICAL TRIAL: NCT05763394
Title: Effects of Polarized Exercise on Cardiovascular Capacity and Lipid Metabolism in Adolescents With Severe Obesity
Brief Title: Effects of Polarized Exercise in Adolescents With Severe Obesity (ALPOLAROB)
Acronym: ALPOLAROB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01C212
Record Dates: First submitted 2023-02-26; First posted 2023-03-10 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Obesity; Exercise Training
Keywords: Obesity; Exercise training; Adolescents; Rehabilitation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polarized workout (Experimental)
  Interventions: Other: Polarized workout program
- High intensity workout (Experimental)
  Interventions: Other: High intensity workout program

INTERVENTIONS:
Other: Polarized workout program — Polarized workout lasting approximately 40 minutes (two sessions/day, 5 days a week), characterized by a 5-minute warm-up performed at 50% of the peak V'O2, followed by 3 sets of 2 minutes at 95% of peak V'O2, interspersed with 1 minute of recovery at 40% of peak V'O2, followed by 30 minutes of moderate activity at 60% of V'O2 peak. Total of 24 sessions in 12 days.
  Arms: Polarized workout
Other: High intensity workout program — High intensity workout (HIIT) (two sessions/day, 5 days a week), characterized by a 10-minute warm-up performed at 50% of peak V'O2 , followed by 6 series of 40 s of high-intensity walking corresponding to 95% of peak V'O2, interspersed with 5 minutes of walking at 40% of peak V'O2, ending with 5' of cool-down at 50% of the peak V'O2. Total of 24 sessions in 12 days.
  Arms: High intensity workout

SUMMARY:
Recent studies have shown that polarized training (i.e. the combination in the same session of intermittent high intensity exercise training, consisting of repeated, short-duration, high-intensity exercises on a cycle ergometer or a treadmill, and moderate exercise) can encourage the participation of obese people in body weight reduction programs, providing more dynamic exercises, less tiring and therefore more acceptable.

To date, no data are available on the effects of polarized exercise in the rehabilitation of obese adolescents, who are often unwilling to engage in prolonged and monotonous motor activities.

The demonstration that the polarized exercise might encourage the participation of obese adolescents in multidisciplinary body weight reduction programs, improve the cardiovascular capacity and also favor an adequate oxidation of lipids during the phase of exercise and post-exercise rest, could support its prescription in the programs of integrated metabolic rehabilitation of adolescent obesity.

DETAILED DESCRIPTION:
Subjects 24 obese adolescents (BMI-standard deviation score > 2), male, age range: 13-18 years, admitted to the Division of Auxology, San Giuseppe Hospital, Istituto Auxologico Italiano, Piancavallo (VB) for a 3-week metabolic rehabilitation program.

Measures:

In basal conditions (hospital admission) and at the end of the metabolic rehabilitation period (21st day), the anthropometric characteristics and body composition will be evaluated by means of tetrapolar impedancemetry (Human-IM Scan, DS-Medigroup, Milan, Italy). In basal conditions all the recruited subjects will undergo an incremental test on a treadmill aimed at determining the maximum lipid oxidation, the peak oxygen consumption value (peak V'O2), and the intensities corresponding to the various percentages of the V' Peak O2 (Medical graphics Corporation, St Paul, MN, USA). Subsequently, subjects will be randomly divided into two groups. The first group (no. 12) will perform a Polarized workout lasting approximately 40 minutes (two sessions/day, 1 in the morning and 1 in the afternoon, 5 days a week), characterized by a 5-minute warm-up performed at 50% of the V 'peak O2, followed by 3 sets of 2 minutes at 95% of peak V'O2, interspersed with 1 minute of recovery at 40% of peak V'O2, followed by 30 minutes of moderate activity at 60% of V'O2 'O2 peak. The second group (no. 12) will perform two sessions (one in the morning and one in the afternoon, 5 days a week) of a high intensity workout (HIIT) characterized by a 10-minute warm-up performed at 50% of peak V'O2 , followed by 6 series of 40 s of high-intensity walking corresponding to 95% of peak V'O2, interspersed with 5 minutes of walking at 40% of peak V'O2, ending with 5' of cool-down at 50% of the peak V'O2. Both workouts (24 sessions in total, spread over 12 days) will be matched for the same calories expended. At the end of the rehabilitation period, all subjects will again be subjected to an incremental test on a conveyor belt with the same execution methods as for the baseline test.

ELIGIBILITY:
Inclusion Criteria:

i. obesity (BMI-standard deviation score > 2) ii. sex: male iii. age range: 13-18 years iv. hospitalization for integrated metabolic rehabilitation program

Exclusion Criteria:

None

Ages: 13 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Peak VO2 | Baseline and at the end of the rehabilitation program (21 days)
  Change in peak VO2

SECONDARY OUTCOMES:
Body fat mass | Baseline and at the end of the rehabilitation program (21 days)
  Change in body fat mass - bioimpedance analysis
Body fat free mass | Baseline and at the end of the rehabilitation program (21 days)
  Change in body fat free mass - bioimpedance analysis
Body weight | Baseline and at the end of the rehabilitation program (21 days)
  Change in body weight
Body mass index | Baseline and at the end of the rehabilitation program (21 days)
  Change in body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Site Piancavallo, Oggebbio, Verbania, Italy